CLINICAL TRIAL: NCT04832113
Title: ETADAPT- Evaluation of the Impact of Patient's Therapeutic Education (PTE) in Adapted Physical Activity (APA) and Dietetic on the Reproducibility of Radiotherapy Sessions for Prostate Cancers.
Brief Title: Impact of Patient's Therapeutic Education in APA and Dietetic on Radiotherapy Reproducibility Sessions for Prostate Cancer
Acronym: ETADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ET20-0284 ETADAPT
Record Dates: First submitted 2021-03-11; First posted 2021-04-05 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Therapeutics Education (PTE) (Experimental): Educational diagnosis prior radiotherapy and participation to Patient Therapeutics Education (PTE) in Adapted Physical Activity (APA) and dietetic sessions. In addition to conventional support (dietary and hydration advice).
  Interventions: Other: Adapted Physical Activity and Dietetic
- Conventional support (Other): Dietary and hydration advices
  Interventions: Other: conventional management

INTERVENTIONS:
Other: Adapted Physical Activity and Dietetic — session in addtion conventional management dietetic, hydratation and physical activity
  Other Names: Follow-up of Adapted Physical Activity and Dietetic Hydratation
  Arms: Patient Therapeutics Education (PTE)
Other: conventional management — Dietary and hydratation advices according to the recommendations
  Other Names: conventional management dietary and hydratation
  Arms: Conventional support

SUMMARY:
The primary objective of this study is to evaluate the impact of Patient's Therapeutic Education (PTE) in Adapted Physical Activity (APA) ans dietetic on the reduction of interventions number on rectal volume (laxative or probe).

The secondary objectives are to evaluate the contribution of Patient's Therapeutic Education (PTE) between the 2 arms on repositionnind during the radiotherapy session, the gastrointestinal toxicity, the need to use laxative or transit regulating treatment or techniques, the quality of life, the undernutrition and food intake, the evolution in eating/hydratation and physical habits.

For the experimetal arm, the satisfaction and the compliance with PTE program will be evaluated, as well as the need of additionnal use of dietary and APA consultations.

DETAILED DESCRIPTION:
Prostate cancer is the 3rd cause of cancer mortality in patient aged over 50 years. Radiotherapy treatment plans require specific conditions:

* Reproductibility of patient's positioning (requiring management of bladder and rectal fillings at each session).
* An image-guided treatment consisting in acquiring an image before each session. This pre-treatment Imaging allows the optimal adjustment of the target volume and organs at risk (bladder and rectum).

To allow reproductibility of target volume positioning at each radiotherapy session, it's recommended to have an empty rectum at the time of the radiotherapy preparation scan, and to check repletion before each session.

It's recommended that the patient has a comfortably full bladder to limit the volume of irradiated bladder mucosa. The radiotherapy teams don't have any recommendations concerning the rectum and manage this problem session by session, according to the repositioning Imaging of the current day.

According to a pilot study carried out in 2017 in the radiotherapy department of the Léon Bérard center, an intervention for a dilated rectum (probe or laxative) was necessary for an average of 25% of session per patient.

These rectal problems can be partly explained by the age (60-80 years) and sedentary lifestyle of patients with prostate cancer. Physical activities, adapted hydratation and changes in eating habits are an integral part of the constipation and flatulence prevention.

ELIGIBILITY:
Inclusion Criteria:

I1: Age >= 18 years old.

I2: Patient with prostatic adenocarcinoma with indication for first-line or post-operative radiotherapy (adjuvant or biologic recurrence).

I3: Patient able to practice a physical activity (certificate of aptitude for adapted physical activity).

I4: Life expectancy greater than 6 months.

I5: Absence of chronic inflammatory intestinal disease or intestinal surgery.

I6: Signed informed consent.

I7: Patient covered by a medical insurance.

I8. At least 20 sessions of radiotherapy planned

Exclusion Criteria:

E1: Patient does not understand and cannot read French.

E2: Patient followed for a psychiatric pathology or presenting cognitive disorders.

E3: Inability to comply with study follow-up goegraphical, social or psychological reasons.

E4: Patient requiring tutorship or curatorship or patient deprived of liberty.

E5: Participation to another clinical trial which may interfere with principal Endpoint assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-06-21 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of Patient's Therapeutic Education in APA on the reduction of interventions number on rectum | An average of 4 months
  Number of uninstallation during the radiotherapy session

SECONDARY OUTCOMES:
Evaluate the contribution of Patient's Therapeutic Education on patient's repositionning efficiency | An average of 4 months
  Rate of patients never uninstalled compared to patients uninstalled during prostate's radiotherapy
Evaluate the contribution of Patient's Therapeutic Education on the gastrointestinal toxicity | An average of 4 months
  Acute gastrointestinal toxicity ≥ grade 2 (NCI- CTCAE V5)
Evaluate the contribution of Patient's Therapeutic Education on the use of laxative or transit regulating treatment or techniques | An average of 4 months
  Prescribed laxatives or transit regulation treatments or techniques
Evaluate the contribution of Patient's Therapeutic Education on patients' quality of life | An average of 4 months
  Using European Organisation for Research and Treatment of Cancer - Core Quality of life questionnaire (QLQC30) (Evaluation of patient's quality of life during the last 7 days - From 4 [worse reply] to 1 [better reply])
Evaluate the contribution of Patient's Therapeutic Education on the undernutrition | An average of 4 months
  Collection of patients' weight (kg)
Evaluate the contribution of Patient's Therapeutic Education on the food intake | An average of 4 months
  Collection of patients' weight (kg)
Evaluate the contribution of Patient's Therapeutic Education on the undernutrition | An average of 4 months
  Using Socio Economic Factor Index scale (SEFI) (Scale from 10 [I ate my entire meal] to 0 [I did not eat anything])
Evaluate the contribution of Patient's Therapeutic Education on the food intake | An average of 4 months
  Using Socio Economic Factor Index scale (SEFI) (Scale from 10 [I ate my entire meal] to 0 [I did not eat anything])
Evaluate the contribution of Patient's Therapeutic Education on the undernutrition | An average of 4 months
  Using the "Eating and hydration habits questionnaire"
Evaluate the contribution of Patient's Therapeutic Education on the food intake | An average of 4 months
  Using the "Eating and hydration habits questionnaire"
Evaluate the contribution of Patient's Therapeutic Education on the evolution in eating habits | An average of 4 months
  Using the "Eating and hydration habits questionnaire"
Evaluate the contribution of Patient's Therapeutic Education on the evolution in hydratation habits | An average of 4 months
  Using the "Eating and hydration habits questionnaire"
Evaluate the contribution of Patient's Therapeutic Education on the evolution in APA habits | An average of 4 months
  Using International Physical Activity Questionnaire (IPAQ) (Description of the physical activity during the last 7 days)
Evaluate patient's satisfaction with Patient's Therapeutic Education program (experimental arm) | An average of 4 months
  Using satisfaction questionnaire (scale from 1 [worse evaluation] to 4 [better evaluation])
Evaluate the compliance to APA session recommendations | An average of 4 months
  Daily collection of steps numbers
Evaluate the compliance to APA session recommendations | An average of 4 months
  Evaluation during phone calls every 15 days
Evaluate the number of patients requiring additional dietetic session | An average of 4 months
  Evaluation during phone calls every 15 days
Evaluate the number of patients requiring additional APA session | An average of 4 months
  Evaluation during phone calls every 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Roux, Principal Investigator — Centre Leon Berard
Locations (5):
- France (5):
  - Chu de saint etienne, Saint-Etienne, Rhône-Alpes Auvergne
  - Groupe Hospitalier Mutualiste de Grenoble Institut Daniel HOLLARD, Grenoble
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain